CLINICAL TRIAL: NCT04635436
Title: Efficacy of Split Gait in the Treatment of Dynamic Asymmetries in Subjects With Pathologic Claudication
Acronym: ESPLICA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Principal Investigator, Luigi Tesio, Prof, MD, Director of the Department of Neuromotor Rehabilitation, Ospedale San Luca, Istituto Auxologico Italiano, IRCCS; Full Professor, Department of Biomedical Sciences for Health, Università degli Studi di Milano, Milan, Italy, Istituto Auxologico Italiano
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 24C902_2019
Record Dates: First submitted 2020-11-13; First posted 2020-11-19 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Multiple Sclerosis; Poststroke/CVA Hemiparesis; Parkinson Disease; Amputation; Knee Impairment
Keywords: walking; split-belt treadmill; motor adaptation; after-effect; dynamic symmetry; rehabilitation
MeSH Terms: conditions — Multiple Sclerosis; Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pathologic group (Other): At least 20 participants with various orthopaedic or neurologic conditions (for example, post-stroke hemiparesis, Parkinson's disease, multiple sclerosis, unilateral amputation, surgical orthopedic interventions) will be enrolled.
  Interventions: Other: Split-belt treadmill walking.

INTERVENTIONS:
Other: Split-belt treadmill walking. — The intervention will consist of split-belt treadmill walking. During the test session, participants will walk on a split-belt treadmill mounted on force sensors with the belts running at the same or at different velocities. They will walk freely without any support. The test sequence will be the following:
  1. Baseline phase. 3 minutes walking at increasing speed, speed will be increased of 0.1 m s-1 every 30 s. A brief pause of around 1 minute will follow.
  2. Habituation phase. 30 seconds walking at 0.2 m s-1.
  3. Adaptation phase. The velocity of the belt under the non-affected lower limb will be increased to 0.6 m s-1, while the other belt will maintain its velocity of 0.2 m s-1 for 6 minutes.
  4. Post-adaptation phase. Belts' velocities will be restored at 0.2 m s-1 for 6 minutes.
  Participants will be informed before the changes in belts' velocities with a verbal warning.
  Participants will repeat the same protocol with the affected lower limb on the fast belt after one week.

SUMMARY:
Walking on a split-belt treadmill (each of the two belts running at a different speed) imposes an asymmetrical gait, mimicking limping that has been observed in various pathologic conditions. This walking modality has been proposed as an experimental paradigm to investigate the flexibility of the neural control of gait and as a form of therapeutic exercise for hemi-paretic patients. However, the scarcity of dynamic investigations both for segmental aspects and for the entire body system, represented by the centre of mass, challenges the validity of the available findings on split gait.

Compared with overground gait in hemiplegia, split gait entails an opposite spatial and dynamic asymmetry. The faster leg mimics the paretic limb temporally, but the unimpaired limb from the spatial and dynamic point of view. These differences suggest that a partial shift in perspective may help to clarify the potential of the split gait as a rehabilitation tool.

The aim of the present study is to investigate the dynamic asymmetries of lower limbs in adults with unilateral motor impairments (e.g. hemiplegia post-stroke, Parkinson's disease, multiple sclerosis, unilateral amputation, surgical orthopedic interventions) during adaptation to gait on a split-belt treadmill. The sagittal power provided by the ankle and the total mechanical energy of the centre of mass will be thoroughly studied. The time course of phenomena both during gait when the belts are running at different speed and when the belts are set back to the same speed (i.e. the after-effect) will be investigated.

A greater dynamic symmetry between the lower limbs is expected after split gait. The question whether this symmetry will occur when the pathological limb is on the faster or the lower belt will be disclosed. Some alterations of the motion of the centre of mass during split gait are also expected.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 70 years old;
* ability to walk for at least 20 meters without support;
* ability to wittingly sign the informed consent form;
* ability to understand the instructions and to complete the motor task;
* visual acuity > 10/20 on the worse side, with optical correction;
* unilateral motor impairments of one lower limb as a consequence of various pathologic conditions, such as (not exhausting list): post-stroke hemiparesis, Parkinson's disease with lateral asymmetry in the motor symptoms, multiple sclerosis with lateral asymmetry in the motor symptoms, unilateral amputation with prosthetic correction, surgical orthopedic interventions, unilateral lesions of peripheral nerves.

Exclusion Criteria:

* systemic neurologic pathologies;
* orthopedic surgical interventions, other than those determining the inclusion criteria;
* symptomatic pathologies of rachis;
* other sensory or neurological pathologies with impact on balance and gait;
* pregnancy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-02-05 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Ankle Joint Power | Two assessments, at one week-interval
  Joint kinematics will be recorded through an optoelectronic method as per the Davis anthropometric model. The 3D displacement of the markers will be captured using 10 near-infrared stroboscopic cameras. Joint power will be computed through the spatiotemporal synchronization of ground reaction force vectors and the joint centers of rotation. Only the sagittal plane will be considered for the analysis. Joint power will be computed as the product of joint torque and joint rotation speed. Power will be defined as positive or generated when the joint moment and rotation speed shared the same directions (i. e., when agonist muscles are contracting while shortening), as negative or absorbed otherwise. Positive work will be computed as the integral of the generated (positive) power over time.

SECONDARY OUTCOMES:
Step Length | Two assessments, at one week-interval
  The sagittal distance between the markers put on the lateral malleolus of the posterior and anterior feet at the ground strike of the anterior foot. The side of step will be defined as the side of the posterior foot during double stance .
Single Stance Time | Two assessments, at one week-interval
  For each lower limb, the time interval during which the limb determines vertical ground reactions equal to or exceeding 30 N.
Double Stance Time | Two assessments, at one week-interval
  The time interval during which, under both lower limbs, vertical ground reactions equal or exceed 30 N. The side of the double stance time will be defined as the side of the posterior foot.
Parameters of the center of mass motion | Two assessments, at one week-interval
  The changes in kinetic energy due to the forward (Ekf), lateral (Ekl) and vertical (Ekv) velocity; the changes of gravitational potential energy (Ep); the changes of the mechanical energy due to the vertical motion, Ev = Ekv+Ep; the changes of the total mechanical energy (Etot = Ekf+Ekl +Ev). The amount of recovery of mechanical energy, R, due to the passive exchange between Ekf, Ev and Ekl, will be calculated according to the equation R = (Wf + Wv + Wl - Wext)/(Wf + Wv + Wl) × 100, where Wf for Ekf, Wv for Ev, Wl for Ekl and Wtot for Etot represents the corresponding work values calculated as the sum of the positive increments of these energy values during one step.

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Tesio, MD, Full professor, Principal Investigator — Istituto Auxologico Italiano
Locations (1):
- Istituto Auxologico Italiano, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Betschart M, Lauziere S, Mieville C, McFadyen BJ, Nadeau S. Changes in lower limb muscle activity after walking on a split-belt treadmill in individuals post-stroke. J Electromyogr Kinesiol. 2017 Feb;32:93-100. doi: 10.1016/j.jelekin.2016.12.007. Epub 2017 Jan 3. PMID 28086163
- [Background] Betschart M, McFadyen BJ, Nadeau S. Repeated split-belt treadmill walking improved gait ability in individuals with chronic stroke: A pilot study. Physiother Theory Pract. 2018 Feb;34(2):81-90. doi: 10.1080/09593985.2017.1375055. Epub 2017 Sep 13. PMID 28901824
- [Background] Helm EE, Reisman DS. The Split-Belt Walking Paradigm: Exploring Motor Learning and Spatiotemporal Asymmetry Poststroke. Phys Med Rehabil Clin N Am. 2015 Nov;26(4):703-13. doi: 10.1016/j.pmr.2015.06.010. Epub 2015 Sep 26. PMID 26522907
- [Background] Lauziere S, Mieville C, Betschart M, Duclos C, Aissaoui R, Nadeau S. Plantarflexion moment is a contributor to step length after-effect following walking on a split-belt treadmill in individuals with stroke and healthy individuals. J Rehabil Med. 2014 Oct;46(9):849-57. doi: 10.2340/16501977-1845. PMID 25074249
- [Background] Malone LA, Bastian AJ. Spatial and temporal asymmetries in gait predict split-belt adaptation behavior in stroke. Neurorehabil Neural Repair. 2014 Mar-Apr;28(3):230-40. doi: 10.1177/1545968313505912. Epub 2013 Nov 15. PMID 24243917
- [Background] Malone LA, Bastian AJ, Torres-Oviedo G. How does the motor system correct for errors in time and space during locomotor adaptation? J Neurophysiol. 2012 Jul;108(2):672-83. doi: 10.1152/jn.00391.2011. Epub 2012 Apr 18. PMID 22514294
- [Background] Reisman DS, Bastian AJ, Morton SM. Neurophysiologic and rehabilitation insights from the split-belt and other locomotor adaptation paradigms. Phys Ther. 2010 Feb;90(2):187-95. doi: 10.2522/ptj.20090073. Epub 2009 Dec 18. PMID 20023001
- [Background] Reisman DS, Block HJ, Bastian AJ. Interlimb coordination during locomotion: what can be adapted and stored? J Neurophysiol. 2005 Oct;94(4):2403-15. doi: 10.1152/jn.00089.2005. Epub 2005 Jun 15. PMID 15958603
- [Background] Reisman DS, McLean H, Keller J, Danks KA, Bastian AJ. Repeated split-belt treadmill training improves poststroke step length asymmetry. Neurorehabil Neural Repair. 2013 Jun;27(5):460-8. doi: 10.1177/1545968312474118. Epub 2013 Feb 7. PMID 23392918
- [Background] Reisman DS, Wityk R, Silver K, Bastian AJ. Locomotor adaptation on a split-belt treadmill can improve walking symmetry post-stroke. Brain. 2007 Jul;130(Pt 7):1861-72. doi: 10.1093/brain/awm035. Epub 2007 Apr 2. PMID 17405765
- [Background] Reisman DS, Wityk R, Silver K, Bastian AJ. Split-belt treadmill adaptation transfers to overground walking in persons poststroke. Neurorehabil Neural Repair. 2009 Sep;23(7):735-44. doi: 10.1177/1545968309332880. Epub 2009 Mar 23. PMID 19307434
- [Background] Selgrade BP, Thajchayapong M, Lee GE, Toney ME, Chang YH. Changes in mechanical work during neural adaptation to asymmetric locomotion. J Exp Biol. 2017 Aug 15;220(Pt 16):2993-3000. doi: 10.1242/jeb.149450. Epub 2017 Jun 8. PMID 28596214
- [Background] Selgrade BP, Toney ME, Chang YH. Two biomechanical strategies for locomotor adaptation to split-belt treadmill walking in subjects with and without transtibial amputation. J Biomech. 2017 Feb 28;53:136-143. doi: 10.1016/j.jbiomech.2017.01.012. Epub 2017 Jan 14. PMID 28126335
- [Background] Tesio L, Malloggi C, Malfitano C, Coccetta CA, Catino L, Rota V. Limping on split-belt treadmills implies opposite kinematic and dynamic lower limb asymmetries. Int J Rehabil Res. 2018 Dec;41(4):304-315. doi: 10.1097/MRR.0000000000000320. PMID 30303831
- [Background] Tesio L, Rota V. Gait analysis on split-belt force treadmills: validation of an instrument. Am J Phys Med Rehabil. 2008 Jul;87(7):515-26. doi: 10.1097/PHM.0b013e31816f17e1. PMID 18388556